CLINICAL TRIAL: NCT02306876
Title: A Randomized,Subject And Investigator Blind, Sponsor Open Placebo Controlled, Parallel Phase 1b Study To Examine The Safety, Pharmacokinetics, And Pharmacodynamic Effects Of Pf-06412562 On Cognitive And Reward/Motivation Domains In Healthy Male Volunteers Selected By Cognitive Phenotype
Brief Title: A Study To Examine Safety, Pharmacokinetics, And Pharmacodynamic Of Pf 06412562 In Healthy Males
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study recruitment was terminated on 14 June 2016 due to a Pfizer business decision. This study was not terminated for reasons of safety.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: B7441004
Record Dates: First submitted 2014-11-20; First posted 2014-12-03 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Healthy
MeSH Terms: interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PF-06412562 3mg (Experimental): PF-06412562 3mg BID
  Interventions: Drug: PF-06412562 3mg BID
- Placebo (Placebo Comparator): Placebo BID
  Interventions: Other: Placebo
- PF-06412562 15mg (Experimental): PF-06412562 15mg BID
  Interventions: Drug: PF-06412562 15mg BID

INTERVENTIONS:
Drug: PF-06412562 3mg BID — PF-06412562
  Other Names: PF-06412562 3mg
  Arms: PF-06412562 3mg
Drug: PF-06412562 15mg BID — PF-06412562
  Other Names: PF-06412562 15mg
  Arms: PF-06412562 15mg
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is designed to investigate the safety, tolerability pharmacokinetics and pharmacodynamic effects of PF-06412562 following multiple dose administration as MR tablets in healthy adult males.

DETAILED DESCRIPTION:
This study is designed to investigate the safety, tolerability pharmacokinetics and pharmacodynamic effects of PF-06412562 following multiple dose administration as MR tablets in healthy adult males. The study will be comprised of 2 analytical stages. Both analytical stages will be conducted as randomized, subject and investigator blind, sponsor open, placebo-controlled, parallel design. Study enrollment will be continuous through Stage I and Stage II. Stage I consists of approximately 45 completer subjects (approximately 15 per arm). Stage I is an exploratory hypothesis generation stage. No multiple comparison adjustment will be conducted for the Stage I analysis. The sample size in Stage I is based on operational feasibility. All endpoints including the composite scores will be tested at the end of Stage I. Each PF-06412562 dose (3 mg BID and 15 mg BID) will be compared to the placebo arm for each endpoint. Up to 5 comparisons that meet Stage I decision criteria will be treated as primary comparisons in Stage II (see Data Analysis section). Stage II is a hypothesis testing stage in which multiple comparisons will be adjusted and overall type I error rate will be controlled across all primary comparisons. Stage II will be formally powered to study those endpoints/doses most likely to demonstrate the strongest pharmacodynamic signal. Stage II will not exceed 56 completers (~21 in each PF-06412562 arm and ~14 in placebo arm). Study enrollment will be continuous through Stage I and Stage II. The three treatments in both stages include (i) PF-06412562 3 mg BID (ii) PF-06412562 15 mg BID, and (iii) placebo. Separate placebo groups, contemporaneous with the treatment groups, will be recruited for Stage I and Stage II. A total of approximately 101 subjects will be randomly assigned to one of the 3 treatments. If a subject drops out before completing the study, or withdraws for reasons unrelated to the safety of the test treatment, the subject will be replaced at the discretion of the Sponsor in consultation with the investigator. Subjects with fMRI or ERP data that does not pass imaging or ERP data QC will also be replaced.

Subjects will be randomized to a specific treatment arm according to the randomization schedule provided to the site by Pfizer. Two doses of PF-06412562 (3 mg and 15 mg), administered as MR tablets, will be given twice daily (BID) from Day 1 through Day 6. A loading dose of PF-06412562 will be administered as an IR tablet on Day 1 only to facilitate rapid attainment of concentration into the target range. For subjects assigned to the 3 mg BID group, one 3 mg MR tablet and one

1 mg PF-06412562 IR tablet will be administered. For subjects assigned to the 15 mg BID group, one 15 mg MR tablet and one 5 mg IR dose of PF-06412562 will be administered.

On Day 7 only the morning dose will be administered. Subject participation will be approximately 12 days (and 11 nights), excluding screening and follow-up. Screening activities will be completed up to 28 days prior to admission to the study on Day -3. The follow-up visit is conducted approximately 7 to 10 days after the last dose of study drug administration. Medically healthy, right-handed male subjects, aged 18-45 will be screened for working memory capacity, psychiatric disorders and other cognitive/educational constrains. Subjects who meet all entry criteria will be randomized into one of the three treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Medically healthy
* Male
* Right-handed aged
* 18-45 years
* BMI 17.5 to 35kg/m2.

Exclusion Criteria:

* Females
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of screening and at the time of dosing).

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 77 (Actual)
Dates: Start 2015-01-19 (Actual); Primary Completion 2016-06-14 (Actual); Study Completion 2016-06-14 (Actual)

PRIMARY OUTCOMES:
change from baseline for Columbia Suicide Severity Rating Scale | Screening, Day 1, Day 7 and Follow-up
  Columbia Suicide Severity Rating Scale

SECONDARY OUTCOMES:
Cavg: Average plasma PF-06412562 and PF-06663872 concentrations at steady state | Day 4, 6 and 8
  Average plasma PF-06412562 and PF-06663872 concentrations for each dose at times 0, 5, and 12 hours on days 4 and 6, as well as 0 hours on Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- United States (3):
  - Arcadia MRI & Imaging Center, Arcadia, California
  - California Clinical Trials Medical Group, Glendale, California
  - Glendale Adventist Medical Center, Glendale, California

REFERENCES:
- [Derived] Balice-Gordon R, Honey GD, Chatham C, Arce E, Duvvuri S, Naylor MG, Liu W, Xie Z, DeMartinis N, Harel BT, Braley GH, Kozak R, Park L, Gray DL. A Neurofunctional Domains Approach to Evaluate D1/D5 Dopamine Receptor Partial Agonism on Cognition and Motivation in Healthy Volunteers With Low Working Memory Capacity. Int J Neuropsychopharmacol. 2020 May 27;23(5):287-299. doi: 10.1093/ijnp/pyaa007. PMID 32055822
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7441004